CLINICAL TRIAL: NCT05610384
Title: Intravenous Ibuprofen Versus Ketorolac for Perioperative Pain Control After Open Hysterectomy: a Randomized Controlled Trial
Brief Title: Ibuprofen Versus Ketorolac for Perioperative Pain Control After Open Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MD-246-2022
Record Dates: First submitted 2022-11-03; First posted 2022-11-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain; Hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketorolac group (Active Comparator): ketorolac 30 mg
  Interventions: Drug: Ketorolac Injectable Solution
- Ibuprofen group (Active Comparator): ibuprofen 800 mg
  Interventions: Drug: Ibuprofen 800 mg

INTERVENTIONS:
Drug: Ketorolac Injectable Solution — ketorolac 30 mg (diluted in 200 mL normal saline) intravenously over 5 minutes before induction of anesthesia then every 8 hours postoperatively
  Arms: Ketorolac group
Drug: Ibuprofen 800 mg — ibuprofen 800 mg intravenously (Diluted in 200 mL of normal saline) over 5 minutes before induction of anesthesia then every 8 hours postoperatively.
  Arms: Ibuprofen group

SUMMARY:
The aim of this study is to compare the analgesic effect of intravenous ibuprofen to ketorolac for pain control after open hysterectomy

DETAILED DESCRIPTION:
Thirty minutes before the surgery, all patients will receive 1 gm paracetamol intravenously then every 6 hours postoperatively.

A research assistant is responsible for opening the envelopes, group assignment and drug preparation (the three doses will be prepared and marked with the patient's name as well as the time of administration) without any further involvement in the study. The patient, attending anesthetist, nurse and data collector will be blinded to the administered drug.

Upon arrival to the operating room, routine monitors (electrocardiogram, pulse oximetry, and non-invasive blood pressure monitor) will be applied; intravenous line will be secured, and prophylactic antiemetic will be provided in the form of slow intravenous injection of 8 mg dexamethasone drugs.

Anesthesia Anesthesia will be induced with 2 mg/kg propofol, 1 mcg/kg fentanyl, and tracheal intubation will be facilitated by 0.5 mg/kg atracurium after loss of consciousness. Anesthesia will be maintained with isoflurane 1-1.2% in oxygen and 0.1 mg/kg atracurium every 20 minutes. Intraoperative analgesia will be in the form of 1 mcg/kg fentanyl boluses as needed.

Postoperatively, pain assessments using the visual analogue scale (VAS) will be performed at rest and during movement (knee flexion) at 0.5, 2, 4, 6, 10, 18, and 24 h after leaving the operating room. If the VAS score is > 3 intravenous titration of 2 mg morphine given slowly to be repeated after 30 minutes if pain persisted.

Intravenous ondansetron 4 mg will be given to treat postoperative nausea or vomiting

ELIGIBILITY:
Inclusion Criteria:

* adult (40-65 years)
* ASA I-II women
* scheduled to undergo open elective abdominal hysterectomy with or without salpingo-oophorectomy

Exclusion Criteria:

* renal impairment,
* allergy to any of study's drugs,
* history of gastrointestinal bleeding or ulceration, or inflammatory bowel disease,
* severe cardiac comorbidity (impaired contractility with ejection fraction < 50%, heart block, significant arrhythmias, tight valvular lesions),
* patients undergoing surgery for suspected gynaecological cancer,
* patients on chronic analgesic medication,
* inability to comprehend the Visual Analogue Pain Scoring Scale

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
mean dynamic VAS | 24 hour after surgery
  average postoperative VAS

SECONDARY OUTCOMES:
static VAS | 30 minutes, 2, 4, 6, 10, 18, 24 hours postoperatively
  a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
dynamic VAS | procedure (during knee flexion)
  a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be')
time to first analgesia requirement | period from extubation until first analgesic requirement during the first 24 hour postoperatively
  hours
morphine consumption | during the first 24 hour postoperatively
  mg
time to independent movement | during the first 24 hour postoperatively
  time from extubation to be able independently mobile e.g. using the bathroom
patients satisfaction | at the end of 24 hour postoperative
  on scale of 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Mohamed Hasanin, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be share upon reasonable request from the PI

REFERENCES:
- [Derived] Amin S, Hasanin A, Attia OA, Mostafa M, Elzayat NS, Elsherbiny M, Eissa AA. Intravenous ibuprofen versus ketorolac for perioperative pain control in open abdominal hysterectomy: a randomized controlled trial. BMC Anesthesiol. 2024 Jun 7;24(1):202. doi: 10.1186/s12871-024-02571-0. PMID 38849734